CLINICAL TRIAL: NCT02301858
Title: Identification of Predictive and Prognostic Markers for Lung Cancer With Metastases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Janna Berg (Other)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Sponsor-Investigator, Janna Berg, Consultant, Sykehuset i Vestfold HF
Organization: Sykehuset i Vestfold HF (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SIV 9743
Record Dates: First submitted 2014-08-04; First posted 2014-11-26 (Estimated); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Lung Cancer; Primary Tumor; Metastases
Keywords: molecular pathology; functional genomics; lung cancer; primary tumor; metastases
MeSH Terms: conditions — Lung Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study arm (Other): Genome analysis of tissue samples.
  Interventions: Genetic: Genome analysis of tissue samples.

INTERVENTIONS:
Genetic: Genome analysis of tissue samples. — Genome analysis of tissue samples.

SUMMARY:
The project aims to compare the histopathological and molecular characteristics of tumour tissue from metastases with similar analyses of the primary tumour in the lung, where it is available.

The investigators will therefore perform analysis of blood samples if possible, to identify predictive markers in blood samples.

DETAILED DESCRIPTION:
The investigators want to make genome analysis of tissue samples. This involves analysing the RNA, DNA methylation, for example in cancer cells. This will provide information regarding somatic changes in cancer cells, such as mutations. All of the investigators analysis will be cancer-focused, with the goal of increasing understanding of the heterogeneity.

The investigators will therefore perform analysis of blood samples if possible, to identify predictive markers in blood samples. This will then be the miRNA, RNA expression or protein expression in blood samples.

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastasizing lung cancer where further treatment is still applicable.

Exclusion Criteria:

* Terminal patients or patients in a reduced general condition with EGOC 3-4, i.e. patients who are confined to bed more than 50% of the day, with no clinical indication to perform sampling of the tumor and metastases.
* Patients where further cancer treatment is no longer applicable.
* Patients with cognitive impairment.
* Patients with inaccessible metastases where sampling may cause distress to the patient and are at increased risk of complications.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-12; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Comparing histopathological and molecular characteristics of tumour tissue from metastases with the primary tumour in the lung | 5 years
  We will do profiling of the mRNA (messenger ribonucleic acid) expression of microRNA and perform single nucleotide polymorphism analysis of cancer tissue and compare the expression using statistical methods such as SAM (Significance analysis and microarrays), PAM (Prediction analysis of microarrays). In addition, we wish to perform specific genetic analysis of cancer-related genes. These will be made with available methods like sequencing or TaqMan assays for specific mutations.
  Blood samples will be analysed by microarray methods for RNA and microRNA in addition to serum analysis of proteins.

CONTACTS AND LOCATIONS:
Locations (1):
- Vestfold Hospital Trust, Tønsberg, Norway